CLINICAL TRIAL: NCT01692145
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group Phase II Study of KCT-0809 in Patients With Dry Eye Syndromes
Brief Title: A Parallel Group Phase II Study of KCT-0809 in Patients With Dry Eye Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KCT1204
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye syndromes; Corneal diseases; Conjunctival diseases
MeSH Terms: conditions — Dry Eye Syndromes; Corneal Diseases; Conjunctival Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KCT-0809 ophtalmic solution (Experimental)
  Interventions: Drug: KCT-0809
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KCT-0809
  Arms: KCT-0809 ophtalmic solution
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KCT-0809 compared to placebo in patients with dry eye syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Corneal and conjunctival damage
* Insufficiency of lacrimal secretion
* Ocular symptom

Exclusion Criteria:

* Severe ophthalmic disorder
* Punctual plugs or surgery for occlusion of the lacrimal puncta

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Score of the Corneal conjunctival staining

CONTACTS AND LOCATIONS:
Locations (1):
- Japan, Tokyo and Other Japanese City, Japan